CLINICAL TRIAL: NCT05144672
Title: Irisin Level in Patients With Diabetic Nephropathy
Brief Title: Irisin And Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer S. Hassan, principal investigator, Assiut University
Other Study IDs: AATHSH
Record Dates: First submitted 2021-11-20; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: Irisin
MeSH Terms: interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: The patient group will include 60 patients with type II DM. They will be subdivided into three groups according to albumin-creatinine ratio ,normoalbuminuric group(less than 30mg/g),which will include 20 patients, microalbuminuric group (ACR =30-300 mg/), which will include 20 patients, and macroalbuminuric group (ACR more than 300mg/g),which will include 20 patients.
  Interventions: Diagnostic Test: Laboratory tests; Other: Estimated glomerular filtration rate (eGFR)
- Control Group: control group will include 30 apparently healthy age-matched and sex-matched individuals.
  Interventions: Other: Anthropometric measurements; Procedure: Electrocardiogram and Fundus examination; Other: Brachial index; Diagnostic Test: Laboratory tests; Radiation: Abdominal ultrasound.

INTERVENTIONS:
Diagnostic Test: Laboratory tests — Fasting blood glucose (FBG), postprandial blood glucose, total cholesterol (CHO), triglycerides (TG), high-density lipoprotein cholesterol and low-density lipoprotein cholesterol (LDL-C), urea, creatinine, and uric acid by point colorimetric assay.
  Serum irisin.
  Groups: Patient Group
Other: Anthropometric measurements — Height, weight, waist circumference, and hip circumference were taken as a way of assessing the nutritional status and BMI
  Groups: Control Group
Procedure: Electrocardiogram and Fundus examination — Fundus examination by direct ophthalmoscope
  Groups: Control Group
Other: Estimated glomerular filtration rate (eGFR) — Estimated glomerular filtration rate (eGFR) was calculated by EPI equation.
  Groups: Patient Group
Other: Brachial index — The ankle-brachial index test compares the blood pressure measured at your ankle with the blood pressure measured at your arm
  Groups: Control Group
Diagnostic Test: Laboratory tests — Glycosylated haemoglobin. ACR,urinary albumin (mg) and creatinine (g).
  Groups: Control Group
Radiation: Abdominal ultrasound. — It will be performed for patients only.
  Groups: Control Group

SUMMARY:
Diabetes mellitus (DM) is a complex, multifactorial, chronic metabolic and endocrine disorder. It has become a threat to global health. It has two types. It is estimated that the number of people with type II will reach 700 million by 2045.

DETAILED DESCRIPTION:
It is associated with acute and chronic complications, acute complications include hypoglycemia, diabetic ketoacidosis, hyperglycemic hyperosmolar state, and hyperglycemic diabetic coma. Chronic complications are further divided into microvascular and macrovascular complications. Chronic microvascular complications are neuropathy, retinopathy, and nephropathy. The later one firstly diagnosed by microalbuminuria. whereas chronic macrovascular complications are coronary artery disease (CAD), peripheral artery disease (PAD), and cerebrovascular disease.

The conventional medications in diabetes treatment, oral and insulin, are focusing on insulin secretion and insulin sensitisation. Oral antidiabetics include, Biguanides, Sulfonylureas, Thiazolidinediones, DPP4 inhibitors, GLP-1 analogue, and SGLT2 inhibitors.

Irisin, a myokin and adipokine secreted by muscles and subcutaneous fat, is an interesting peptide performing significant functions in human health. Irisin has been linked to human obesity and insulin resistance status.

Irisin is involved in regulating the mitochondrial function of muscle cells, so increases energy consumption of the body, promotes metabolism and reduces body weight so improves insulin sensetivity. In our study we aim to clarify the effect of antidiabetics on serum irisin in patients with typeII DM who developed diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

Any patients above 40 years with type 2 diabetes of at least two years duration complicated with diabetic nephropathy.

Exclusion Criteria:

* Patients below 40 yrs.
* Patients with type 1 diabetes complicated with diabetic nephropathy
* Type2 diabetes without nephropathy.
* Diabetic nephropathy cases on dialysis due to other causes
* Blood pressure more than 160/100
* Acute coronary syndrome in the past 6 months
* Non alcoholic fatty liver disease, impaired liver function.
* Malignancy.
* Pregnancy
* Acute infection, acute inflammation.
* Severe renal impairment, and urinary tract infection.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients above 40 years with type 2 diabetes of at least two years duration complicated with diabetic nephropathy.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The relation between different stages of diabetic nephropathy and irisin level. | 1 year
  measurement of irisin level in patients with diabetic nephropathy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xuan X, Lin J, Zhang Y, Zhou L, Xu L, Jia J, Zhao B, Lin Z, Zhu Q, Li L, Wu T, Zhang S, Jiang H, Wang Y. Serum Irisin Levels and Clinical Implication in Elderly Patients With Type 2 Diabetes Mellitus. J Clin Med Res. 2020 Sep;12(9):612-617. doi: 10.14740/jocmr4261. Epub 2020 Aug 15. PMID 32849950
- [Background] Ravaut M, Sadeghi H, Leung KK, Volkovs M, Kornas K, Harish V, Watson T, Lewis GF, Weisman A, Poutanen T, Rosella L. Predicting adverse outcomes due to diabetes complications with machine learning using administrative health data. NPJ Digit Med. 2021 Feb 12;4(1):24. doi: 10.1038/s41746-021-00394-8. PMID 33580109
- [Background] Tan SY, Mei Wong JL, Sim YJ, Wong SS, Mohamed Elhassan SA, Tan SH, Ling Lim GP, Rong Tay NW, Annan NC, Bhattamisra SK, Candasamy M. Type 1 and 2 diabetes mellitus: A review on current treatment approach and gene therapy as potential intervention. Diabetes Metab Syndr. 2019 Jan-Feb;13(1):364-372. doi: 10.1016/j.dsx.2018.10.008. Epub 2018 Oct 10. PMID 30641727